CLINICAL TRIAL: NCT01759160
Title: Hemodynamic Responses During Induction: Comparison of Marsh and Schnider Pharmacokinetic Models in Propofol Plasma Target-controlled Infusion
Brief Title: Hemodynamic Responses During Induction: Comparison of Marsh and Schnider Pharmacokinetic Models
Acronym: TCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xia Feng, Department of Anesthesiology, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NSFCfengxiar1; Fengxia1 (Other Grant/Funding Number: NSFC3140050)
Record Dates: First submitted 2012-12-20; First posted 2013-01-03 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Target control infusion; propofol; cardiac depression; induction of anesthesia; hemodynamics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Marsh (Active Comparator): Marsh Plasma TCI with high initial target
  Interventions: Procedure: Marsh Plasma TCI with high initial target
- Schnider (Active Comparator): Schnider Plasma TCI with high initial target
  Interventions: Procedure: Schnider Plasma TCI with high initial target

INTERVENTIONS:
Procedure: Marsh Plasma TCI with high initial target — plasma target-controlled infusion in Marsh model(n=30) with an initial target concentration of 4 μg/ml. Target was then reset and gradually titrated to a sedation level with narcotrend index below 64.
  Other Names: Plasma target-controlled infusion in Marsh model
  Arms: Marsh
Procedure: Schnider Plasma TCI with high initial target — plasma target-controlled infusion in Schnider model(n=30) with an initial target concentration of 4 μg/ml. Target was then reset and gradually titrated to a sedation level with narcotrend index below 64.
  Other Names: Plasma target-controlled infusion in Schnider model
  Arms: Schnider

SUMMARY:
To compare the hemodynamic changes during anesthesia induction between Marsh and Schnider plasma TCI models. We put forward a hypothesis that, if one TCI model is associated with much more prominent vasodilation effect or cardiac depression, a more sharp decrease in mean arterial pressure, systemic vascular resistance , central venous return or stroke volume would be observed.

DETAILED DESCRIPTION:
Current systems of propofol TCI are pre-programmed with the Marsh and Schnider pharmacokinetic models. Rate constants of Marsh are fixed, whereas compartment volumes and clearances are weight proportional. Schnider model has fixed values for VC, V3, k13, and k31, adjusts V2, k12, and k21 for age, and adjusts k10 according to total weight, lean body mass (LBM), and height. One major beneﬁt of the Schnider model is that it adjusts doses and infusion rates according to patient age. This provides a strong argument for using the Schnider model in the elderly and unwell patients which may improve hemodynamic stability and safety.

However for the vast majority of young and middle age patients, whether Marsh or Schnider would be a better choice for hemodynamic stability remains unknown.

With marsh model, as VC is scaled to body weight, the amount of drug delivered is dependent of body weight. In the Schnider model, as VC at 4.27L is independent of body weight, VC in terms of ml/kg decreases as body weight increases. This and the influence of height and weight on clearance results in heavier patients receiving less propofol on a mg/kg basis whereas those with a lower lean body mass will initially receive about 30% less than delivered by Marsh, but after 30 min, the Schnider model delivers about 15% more. Besides, when Schnider model is used in the morbidly obese, the LBM equation can generate paradoxical values resulting in excessive increases in maintenance infusion rates. Nevertheless, the purpose of this study was to investigate the vast majority of Asian patients whose body weight were in normal range. Only patients with BMI between 18 and 29 were included to minimize the influential factor of body weight in TCI system.

To compare the hemodynamic changes during anesthesia induction between Marsh and Schnider plasma TCI models. We put forward a hypothesis that, if one TCI model is associated with much more prominent vasodilation effect or cardiac depression, a more sharp decrease in mean arterial pressure, systemic vascular resistance , central venous return or stroke volume would be observed.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 years and 70 years
* ASA physical status I and II
* surgical procedures requiring general anesthesia with continuous CVP and arterial pressure monitoring.

Exclusion Criteria:

* Patients younger than 16 y or older than 65 y
* Body Mass Index (BMI) <18 or >30
* emergency surgery
* allergy to any of the drugs used
* inability to communicate effectively
* severe cardiovascular dysfunction
* patient refusal and patients on long-term opioids or sedative medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xia Feng, M.D., Principal Investigator — The First Affiliaed Hospital of Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang XY, Zhou ZB, Yang L, Zhou X, Niu LJ, Feng X. Hemodynamic responses during induction: comparison of Marsh and Schnider pharmacokinetic models. Int J Clin Pharmacol Ther. 2015 Jan;53(1):32-40. doi: 10.5414/CP202141. PMID 25500489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process started from Dec. 2012, ended in Jan.2013. Study location is The First Affiliated Hospital of Sun Yat-sen University.
Pre-assignment Details: enrolled participants were excluded when they were found allergic to drugs used during the study.
Groups:
- Marsh: Plasma TCI in Marsh Model with an initial target of 4 μg/ml, gradually titrated according to sedation level.
- Schnider: Plasma TCI in Schnider Model with an initial target of 4 μg/ml, gradually titrated according to sedation level.
Period: Overall Study
Arm/Group | Marsh | Schnider
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marsh | Schnider | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.1) | 41.6 (10.6) | 40.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: SVI (Stroke Volume Index) Value Change From Baseline Level at the End of the First 25 Minutes.
Description: After propofol infusion started, according to sedation level, TCI targets were gradually titrated to reach a state of equilibrium at the end of the first 25 minutes. SVI were continuously monitored, at the end of the first 25 minutes, value change from baseline level were calculated.
Time Frame: The end of the first 25 minutes after propofol infusion
Measure: Mean (Standard Deviation); unit: ml/beat/m^2
Arm/Group | Marsh | Schnider
Number analyzed (Participants) | 30 | 30
ml/beat/m^2 | -31.1 (9.8) | -31.7 (9.9)

2. Secondary Outcome: NI (Narcotrend Index) Reduction
Description: Narcotrend was utilized to continuously record patients' sedation level during induction, provided as a criteria for Cpt (Plasma Target Concentration) adjustment.
Time Frame: 25 minutes after propofol infusion
Reporting Status: Not Posted

3. Secondary Outcome: CVP (Central Venous Pressure)
Description: CVP was continuously monitored to assess preload condition and served to calculate SVRI (systemic vascular resistance index) every minute during the first 25 minutes of infusion.
Time Frame: 25 minutes after induction
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Marsh | Schnider
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marsh (N=30) | Schnider (N=30)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marsh (N=30) | Schnider (N=30)
Hypotension (Systolic blood pressure lower than 75mmHg) (Cardiac disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No